CLINICAL TRIAL: NCT03271203
Title: Patient Interviews to Better Understand Disease Experience and Unmet Treatment Needs in Hand Osteoarthritis
Brief Title: Subject Insights to Understand the Hand Osteoarthritis (HOA)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 206599
Record Dates: First submitted 2017-06-29; First posted 2017-09-05 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis
Keywords: Michigan Hand Outcomes Questionnaire; Real-time data capture; Cognitive debriefing; Hand Osteoarthritis; Concept elicitation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects participating in the CE and CD interview: Thirty adult subjects from the US with erosive HOA will be asked to participate in CE and CD interviews.
  Interventions: Other: Michigan Hand Outcomes Questionnaire
- Subjects participating in interview and real time data capture: Ten adult subjects from the US (n=5 with erosive HOA, n=5 with non-erosive HOA) of the thirty subjects who are participating in the CE and CD interviews, will be asked to participate in the real-time data capture app task
  Interventions: Other: Michigan Hand Outcomes Questionnaire; Other: Real-time data capture app

INTERVENTIONS:
Other: Michigan Hand Outcomes Questionnaire — The MHQ is a self-report measure that assesses the function of the hand(s) and/or wrist(s). The MHQ contains six distinct scales including overall hand function, activities of daily living, pain, work performance, aesthetics and subject satisfaction with hand function. In the pain scale, high scores indicate greater pain, while in the other five scales, high scores denote better hand performance.
Other: Real-time data capture app — Real time data capture app is a smart-phone or web-based application which will allow the subjects to provide responses about their experience of HOA in real-time via varying video, audio, photographic and text forms.
  Groups: Subjects participating in interview and real time data capture

SUMMARY:
Osteoarthritis (OA) is a degenerative joint disease which causes joints to become painful and stiff. HOA is the second most common form of OA and is characterized by stiffness, joint pain and inflammation and tenderness in the knuckles or around the waist. This cross-sectional, qualitative interview study aims to explore the experience of erosive HOA as well as explore the content validity of the Michigan Hand Outcomes Questionnaire (MHQ) by conducting semi-structured combined concept elicitation (CE) and cognitive debriefing (CD) telephone interviews and real-time data capture. The conceptual model developed from this data will be used to support the development of GSK3196165, a human monoclonal antibody target for the treatment of HOA. The CE interviews (45 minutes duration) will explore the experience of subjects suffering with HOA and will collect information about symptoms, health related quality of life (HRQoL), treatment experience and the language used by subjects to describe them whereas the CD interviews (45 minutes duration) will assess the content validity of the MHQ. The real-time disease experience of subjects will be captured by the real-time data capture app-based activity over a period of 7 days. Approximately 30 subjects from the United States (US) of which 15 subjects will be erosive HOA and rest 15 will be non-erosive HOA.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Erosive Hand OA

* Subject is a male or female between 40-80 years of age (inclusive) at the time of signing the informed consent form.
* Subject meets the American College of Rheumatology (ACR) classification of osteoarthritis: Hand pain, aching, or stiffness and 3 or 4 of the following features: Hard tissue enlargement of 2 or more of 10 selected joints, Hard tissue enlargement of 2 or more distal interphalangeal (DIP) joints, Fewer than 3 swollen metatarsophalangeal (MCP) joints or Deformity of at least 1of 10 selected joints where The 10 selected joints are the second and third DIP, the second and third proximal interphalangeal (PIP), and the first carpometacarpal joints of both hands.
* Subject has erosive disease on at least 1 PIP or 1DIP joint as demonstrated by imaging evidence [can include X-ray, ultrasound or magnetic resonance imaging (MRI) evidence].
* Subject has active disease in at least one hand, with at least two soft tissue swollen and tender PIP and/or DIP joints in the affected hand by clinical examination within the past 3 months. If only one hand is affected by HOA and meets the inclusion criteria, the affected hand should be documented at screening and used for all assessments. In cases where both hands are affected by HOA and both meet the inclusion criteria, then the dominant hand should be documented at screening and used for all assessments.
* Subject's self-reported average hand-pain intensity over the past 7 days must be at least '4' on a 0-10 Numerical Rating Scale (NRS).
* Subject must have negative titer rheumatoid factor (RF) and anti- Cyclic Citrullinated Peptide (CCP) antibody.
* Subject must have a personally signed and dated written informed consent form prior to admission to the study.
* Subject must be verbally fluent and literate in English.
* Subject must be able to attend and participate in two 45 minute telephone or video call (Skype or Facetime) interviews (either on the same day or separate days).

Inclusion Criteria for Non-Erosive Hand OA

* Subject is a male or female between 40-80 years of age (inclusive) at the time of signing the informed consent form
* Subject meets the American College of Rheumatology (ACR) classification of osteoarthritis: Hand pain, aching, or stiffness and 3 or 4 of the following features: Hard tissue enlargement of 2 or more of 10 selected joints, Hard tissue enlargement of 2 or more distal interphalangeal (DIP) joints, Fewer than 3 swollen metacarpophalangeal (MCP) joints, Deformity of at least 1 of 10 selected joints where the 10 selected joints are the second and third distal interphalangeal (DIP), the second and third proximal interphalangeal, and the first carpometacarpal joints of both hands.
* Subject has at least 1 finger joint (DIP or PIP) with K-L ≥ 2 [by x-ray in last 12m]. Participant's self-reported average hand-pain intensity over the past 7 days must be moderate to severe (≥4 on a 0-10 Numeric Rating Scale [NRS] or ≥40mm on a 0-100mm Visual Analog Scale [VAS]). If only one hand is affected by hand osteoarthritis (HOA) and meets the inclusion criteria, the affected hand should be documented at screening and used for all assessments. In cases where both hands are affected by HOA and both meet the inclusion criteria, then the dominant hand should be documented at screening and used for all assessments.
* Subject is unwilling or unable to take non-opiate analgesics, or is inadequately controlled by non-opiate analgesics (non-opiate analgesics include Tramadol)
* Subject must have negative titer rheumatoid factor (RF) and anti-CCP antibody
* Subject must have a personally signed and dated written informed consent form prior to admission to the study
* Subject must be verbally fluent and literate in English
* Subject must be able to attend and participate in two 45 minute telephone or video call (Skype or Facetime) interviews (either on the same day or separate days)

Inclusion criteria for subjects taking part in real-time data capture:

* Subject owns/or has access to either a smartphone [iPhone Operating System (iOS) or android] or tablet which has video, audio/microphone and photographic capabilities and access to either the Apple app store or Google play store to download the app.
* Subject is willing and able to take part in the real time data application task and respond to a series of questions/tasks fielded via the application over the course of seven days.]
* Subject would feel comfortable recording short videos of themselves and providing audio commentary in response to app questions/tasks.

Exclusion Criteria:

Exclusion Criteria for Erosive Hand OA

* Subject has history of any clinically significant inflammatory disease other than inflammatory osteoarthritis, especially, but not limited to, rheumatoid arthritis or spondylarthropathies.
* Subject has a diagnosis of rheumatoid arthritis, fibromyalgia, gout, calcium pyrophosphate deposition disease (CPPD), pseudogout, hemochromatosis or other inflammatory rheumatological or autoimmune disorders.
* Subject has had a clinical suspicion of, or previous investigation for CPPD or pseudogout, or history of chondrocalcinosis.
* Subject has any injury, medical or surgical procedure to the affected joint(s) that may interfere with evaluation of the target hand osteoarthritis joint(s).
* Subject has great difficulty hearing, reading or speaking.
* Subject has an uncontrolled psychiatric condition (example, schizophrenia,bipolar disorder) or mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study or likely to have difficulty participating in two 45 minute interviews.
* Subject has severe physical, neurological or cognitive deficits that might prohibit the ability to participate in an interview about the experience of their hand osteoarthritis and completion of a questionnaire.
* Subject is currently or has previously been enrolled in a clinical trial for OA in the past 6 months.

Exclusion Criteria for Non-Erosive Hand OA

* Subject has erosive disease on any proximal interphalangeal (PIP) or distal interphalangeal (DIP) joints as evidenced via X-ray, MRI or ultrasound
* Subject has history of any clinically significant inflammatory disease other than inflammatory osteoarthritis, especially, but not limited to, rheumatoid arthritis or spondylarthropathies
* Subject has a diagnosis of rheumatoid arthritis, fibromyalgia, gout, calcium pyrophosphate deposition disease (CPPD), pseudogout, hemochromatosis or other inflammatory rheumatological or autoimmune disorders
* Subject has had a clinical suspicion of, or previous investigation for CPPD or pseudogout, or history of chondrocalcinosis
* Subject has any injury, medical or surgical procedure to the affected joint(s) that may interfere with evaluation of the target hand osteoarthritis joint(s)
* Subject has great difficulty hearing, reading or speaking
* Subject has an uncontrolled psychiatric condition (e.g., schizophrenia, bipolar disorder) or mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study or likely to have difficulty participating in two 45 minute interviews
* Subject has severe physical, neurological or cognitive deficits that might prohibit the ability to participate in an interview about the experience of their hand osteoarthritis and completion of a questionnaire
* Subject is currently or has previously been enrolled in a clinical trial for hand OA in the past six months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty adult US-English speaking subjects with erosive HOA will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with hand osteoarthritis participating in CE interviews | 1 day
  CE interviews will be carried out to explore disease experience with respect to symptoms, impacts and treatment/surgical experiences.

SECONDARY OUTCOMES:
Content validity of the Michigan Hand Outcomes Questionnaire through CD interviews | 1 day
  The MHQ is a self-report measure that assesses the function of hand(s) and/or wrist(s). The MHQ contains six distinct scales including overall hand function, activities of daily living, pain, work performance, aesthetics and subject satisfaction with hand function. In a pain scale, high scores indicate greater pain, while in the other five scales, high scores denote better hand performance. Subjects will be asked to complete the MHQ questionnaire during CD interview using a 'think-aloud' technique to evaluate the content validity.
Analysis of hand osteoarthritis experience by using real-time data data capture task | Up to 7 days
  A subgroup of ten of the thirty subjects participating in the CE and CD interviews will be asked to take part in the real-time data capture task over the course of 7 days and during this time a series of questions/tasks will be asked to subjects via the application to explore the experience of the symptoms, HRQoL impacts and treatment of erosive HOA and any day-to-day variability that exists these experiences in 'real time'.
Preparation of conceptual model | Up to 7 days
  Data obtained from the CE and CD interviews as well as real-time data capture will be used to develop a conceptual model for erosive HOA. Symptom, impact, and treatment concepts which have been identified will be grouped into domains and displayed visually and any identified relationships or trends between domains will also be included in the model. A key will be developed using color coding or bolding/italics to show the source of the concept (example, red if the concept emerged from the interviews only, and green it emerged from the real-time data capture only). In addition, and where relevant the frequency at which a concept was reported across sources will be included in the model.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bollington, Cheshire, United Kingdom

REFERENCES:
- See also: Results for study 206599 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/206599?search=study&study_ids=206599#rs